CLINICAL TRIAL: NCT03064958
Title: The Postprandial Effects of a High Fat Meal Containing Spices on Endothelial Function: a Pilot Study
Brief Title: The Acute Effect of Spices on Vascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: McCormick Science Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PKE SPICE PILOT
Record Dates: First submitted 2016-09-14; First posted 2017-02-27 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Oxidative Stress
Keywords: glucose regulation; lipids; Immune markers; Endothelium, Vascular
MeSH Terms: interventions — Spices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): Consumption of a high fat meal (1000kcal, 45g fat)
  Interventions: Other: High fat meal
- Spice 2g (Experimental): Consumption of a high fat meal (1000kcal, 45g fat) with 2g of spice (mix of black pepper, basil, bay leaf, cinnamon, coriander, cumin, ginger, oregano, parsley, rosemary, red pepper, turmeric and thyme) incorporated into the meal.
  Interventions: Other: Herbs and spices; Other: High fat meal
- Spice 6g (Experimental): Consumption of a high fat meal (1000kcal, 45g fat) with 6g of spice (mix of black pepper, basil, bay leaf, cinnamon, coriander, cumin, ginger, oregano, parsley, rosemary, red pepper, turmeric and thyme) incorporated into the meal.
  Interventions: Other: Herbs and spices; Other: High fat meal

INTERVENTIONS:
Other: Herbs and spices — Mix of commonly used herbs and spices
  Arms: Spice 2g; Spice 6g
Other: High fat meal — Meal containing 1000kcal and 45g fat

SUMMARY:
The investigators aim to conduct a 3-period randomized controlled crossover study to investigate the postprandial effects of a high fat meal with spice on endothelial function, lipids/lipoproteins, immune function and plasma markers of antioxidants and oxidative stress. Metabolomic profiling will also be conducted. In random order, participants will consume either a high fat meal (1000kcal, 45g fat) or a high fat meal containing 2g of spice or a high fat meal containing 6g of spice. Between each treatment there will be a washout period of at least 3 days. It is hypothesized that consumption of a high fat meal with spice will attenuate postprandial endothelial impairment and triglyceride levels in a dose response manner compared with a high fat meal.

DETAILED DESCRIPTION:
A 3-period randomized controlled crossover study will be conducted to investigate the postprandial effects of a high fat meal with spices on endothelial function, lipids/lipoproteins, immune function, plasma antioxidants and markers of oxidative stress. Metabolomic profiling will also be conducted. In random order participants will consume either a high fat meal (1000kcal, 45g fat) or a high fat meal containing 2g of spices or a high fat meal containing 6g of spices with a 3 day washout period between each treatment. The following spices will be incorporated into the meal black pepper, basil, bay leaf, cinnamon, coriander, cumin, ginger, oregano, parsley, rosemary, red pepper, turmeric and thyme.

Endothelial function will be measured by flow mediated dilation of the brachial artery in the fasting state and 2 and 4 hours after the meal. Participants will also provide a fasting blood sample and samples will also be taken at 1, 2, 3 and 4 hours after the meal.

ELIGIBILITY:
Inclusion Criteria:

* male aged 40-65 years
* BMI 25-35kg/m2
* nonsmoking
* waist circumference =/> 94cm and at least one other CVD risk factor (elevated LDL-C (> 130 mg/dL), CRP (> 1 mg/L), elevated Triglycerides (≥ 150 mg/dL), reduced HDL-cholesterol (< 40 mg/dL), elevated blood pressure (systolic BP ≥ 130 or diastolic BP ≥ 85 mm Hg), elevated fasting glucose (≥ 100 mg/dL))
* low herb/spice consumers (consumption <1/day)

Exclusion Criteria:

* Chronic disease risk factors that are diagnostic of diabetes (fasting glucose > 126 mg/dL) or hypertension (SBP >160 mm Hg or DBP > 100 mm Hg).
* Prescription of anti-hypertensive or glucose lowering drugs.
* Established CVD, stroke, diabetes, liver, kidney or autoimmune disease
* Use of cholesterol/lipid-lowering medication or supplements (psyllium, fish oil, soy lecithin, and phytoestrogens) and botanicals
* weight loss of ≥10% of body weight within the 6 months prior to enrolling in the study
* vegetarianism

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Change in endothelial function measured by flow mediated dilation (FMD) of the brachial artery | Change from baseline at 2 hours and 4 hours after meal consumption

SECONDARY OUTCOMES:
Lipids and lipoproteins | Change from baseline during the 4 hours after meal consumption
Plasma Inflammatory cytokines | Change from baseline during the 4 hours after meal consumption
Inflammatory cytokines in isolated peripheral blood mononuclear cells | Change from baseline during the 4 hours after meal consumption
Glucose | Change from baseline during the 4 hours after meal consumption
Insulin | Change from baseline during the 4 hours after meal consumption
Plasma antioxidants (hydrophilic ORAC, lipophilic ORAC, total ORAC) | Change from baseline during the 4 hours after meal consumption
Oxidative stress | Change from baseline during the 4 hours after meal consumption
Plasma nitrite and nitrate | Change from baseline during the 4 hours after meal consumption
Plasma and Urine Metabolomic profiling | Change from baseline during the 4 hours after meal consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oh ES, Petersen KS, Kris-Etherton PM, Rogers CJ. Spices in a High-Saturated-Fat, High-Carbohydrate Meal Reduce Postprandial Proinflammatory Cytokine Secretion in Men with Overweight or Obesity: A 3-Period, Crossover, Randomized Controlled Trial. J Nutr. 2020 Jun 1;150(6):1600-1609. doi: 10.1093/jn/nxaa063. PMID 32211803